CLINICAL TRIAL: NCT05887089
Title: Verification of the Absence of Analytical Impact of the Transport of Pathological Biological Material by Drone Within the Amiens-Picardie University Hospital
Brief Title: Analytical Impact of the Transport of Pathological Biological Material by Drone
Acronym: PATH-AIRCHU
Status: Withdrawn | Type: Observational
Why Stopped: no participants enrolled
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2023_843_0030
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Biological Samples
Keywords: drone transport; biological samples; unmanned aerial system; UAS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — One supernumerary tube of blood sample for biochemistry analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- no intervention
- drone transportation
  Interventions: Other: drone transport

INTERVENTIONS:
Other: drone transport — additional transport of samples at room temperature by drone (departure from the CHU Amiens-Picardie, 1 hour flight in the CHU Amiens-Picardie air perimeter, return to the CHU Amiens-Picardie)
  Groups: drone transportation

SUMMARY:
The Hospital Group of Territory Somme Littoral Sud, through its biology sector and in partnership with the company DELIVRONE, aims to engage in the experiment of transporting biological samples by means of a drone platform. Transport by air will be between the CHAM, the Abbeville Hospital and the CHU Amiens-Picardie by flying as much as possible over the waterways via the Somme. With a flight speed of around 100km/h at an altitude between 80 and 120 m, drones will be able to connect sites in less than an hour by transporting packages between 2 and 3 kg. Powered by propellers connected to rechargeable batteries, these drones do not emit CO2. This type of transport has not been validated in France by measuring the analytical impact of transport constraints for medical biology, and has never been evaluated according to the criteria of ISO 15189 standard allowing the certification of medical biology laboratories. Validation steps of this transportation method are therefore necessary on pathological samples prior to routine use. The aim of the project is to verify the absence of analytical impact of the transport of pathological biological samples by drone under defined flight conditions, according to the ISO15189 norm.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Amiens-Picardie University Hospital and having benefited from medical biology examinations including the parameters of interest
* according to the usual management modalities and without additional sampling
* at the time of the test period

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: If eligible for the study, patients from the central blood collection unit and the day hospitals of the CHU Amiens-Picardie will be offered to participate in the study. After information and consent of the patient, blood sampling will be performed to obtain the samples necessary for the normal medical management of the patient, as well as additional tubes corresponding to the same prescribed analyses. The collection of the extra tubes will therefore be done at the same time as the routine collection, without any additional invasive procedure.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
variation of ASAT concentration between both groups | one day
variation of ALAT concentration between both groups | one day
variation of BNP concentration between both groups | one day
variation of LDH concentration between both groups | one day
variation of Glucose concentration between both groups | one day
variation of Troponin concentration between both groups | one day
variation of Potassium concentration between both groups | one day
variation of HIL concentration between both groups | one day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No